CLINICAL TRIAL: NCT00443781
Title: Study Of Disc Anaesthesia For The Preoperative Diagnosis Of Chronic Lower Back Pain
Acronym: SODA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Spine LLC (Industry)
Responsible Party: Sponsor
Organization: Medtronic Spinal and Biologics (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SP0603
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Results first posted 2010-08-23 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2012-03

CONDITIONS: Low Back Pain
Keywords: low back pain, degenerative disc disease
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PD and F.A.D. diagnostic testing (Other)
  Interventions: Procedure: functional anesthetic discography; Procedure: provocative discography

INTERVENTIONS:
Procedure: functional anesthetic discography — Functional Anesthetic Discography (F.A.D.) involves the placement and anchoring of a small catheter into a disc. After placement, functional testing is performed, in which the subject elicits his/her back pain via functional maneuvers or postures. Local anaesthetic is then delivered into the target disc through the catheter and the effect on functional back pain is noted.
Procedure: provocative discography — Provocative discography (PD) has been used as a preoperative diagnostic tool for patients with back pain attributed to degenerative disc disease considering lumbar disc surgery. During PD, a clinically suspected disc is accessed with a needle and injected under pressure with radiopaque contrast dye. The subject rates his/her experience of pain for intensity and whether the pain is exactly the same as ("concordant") or different from ("not concordant" or "discordant") typical back pain.

SUMMARY:
The primary objective of this study is to document and compare diagnostic test results and procedure safety in subjects undergoing both Functional Anaesthetic DiscographyTM (F.A.D.) and provocative discography (PD) and determine the appropriateness of the F.A.D. procedure data collection script for use in a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21.
* Chronic axial low back pain without radicular pain for > six months, not responding to at least three months of non-surgical management under the direction of a physician.
* One or two discs at L5/S1, L4/L5 or L3/L4 with abnormal findings by MRI, including any of the following: loss of disc hydration, loss of disc height, high intensity zone (HIZ), Modic changes at adjacent vertebral endplates, or herniation without nerve root compression.
* Subject states that he/she is willing to undergo lumbar spinal fusion, disc replacement, or other definitive treatment if eventual diagnosis supports such treatment.
* Physician believes that discography is clinically indicated for the purpose of surgical decision-making for the subject.
* Pre-treatment low back pain by numerical rating scale (NRS) score > 4 (measured as average in last 24 hours on a 0-10 scale).
* Pre-treatment Oswestry Disability Index (ODI) > 40 (0 - 100 scale).
* Subject states availability for all study visits.
* Subject is able to understand the risks and benefits of participating in the study and provides written informed consent.

Exclusion Criteria:

* Known osteoporosis or osteopenia, metabolic bone disorder, or history of chronic steroid use (the equivalent of 7.5 milligrams of daily prednisone use for > 6 months).
* Suspected painful disc degeneration (based on clinical examination and MRI findings) outside of L5/S1, L4/L5 or L3/L4 levels.
* MRI shows disc abnormalities (listed in Inclusion Criteria #3) at all 3 lower lumbar discs (L3/L4, L4/L5 and L5/S1).
* Abnormal neurologic exam attributable to lumbar disc disease, herniation, or lumbar stenosis.
* Back, buttock or pelvic pain suspected to be due to spinal stenosis, spinal fractures, infection, cancer, facet arthropathy or other hip or pelvis pathology.
* Schmorl's node or endplate disruption evident on MRI at L5/S1, L4/L5, or L3/L4.
* Medical history, physical examination or radiographic evidence (e.g., disc height too narrow) to suggest that either PD or F.A.D. may not be technically feasible.
* Any previous lumbar spine fusion or disc replacement.
* More than grade 1 spondylolisthesis as assessed by x-ray or MRI.
* Significant clinical comorbidity that may potentially interfere with data collection or follow-up (e.g., dementia, severe comorbid illness).
* History of major depression, psychosis or somatization disorder, or panic disorder.
* Allergy to any materials used in PD or F.A.D. devices, contrast, lidocaine, or bupivacaine.
* Any evidence of disc or systemic infection.
* Pregnant or child-bearing potential and not currently on adequate birth control method.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ray M Baker, MD, Principal Investigator — University of Washington; Rick D Guyer, MD, Principal Investigator — Texas Back Institute, Plano, TX
Locations (10):
- United States (10):
  - The Spine and Neurosurgery Center, Huntsville, Alabama
  - Spine Source, Beverly Hills, California
  - Pacific Spine Clinic, Escondido, California
  - UCSD Orthopaedic Surgery, San Diego, California
  - Emory Orthopaedics & Spine Center, Atlanta, Georgia
  - Hanover Orthopaedic Associates, Inc., Hanover, Pennsylvania
  - Texas Back Institute, Plano, Texas
  - East Texas Medical Center, Tyler, Texas
  - Evergreen Surgical Center, Kirkland, Washington
  - Milwaukee Neurological Institute, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- PD and F.A.D. Diagnostic Testing: Subjects with chronic axial low back pain with suspected degenerative disc disease underwent provocative discography(PD)followed by Functional Anaesthetic Discography (F.A.D.)as part of a pilot, multicenter, prospective, single-arm diagnostic study.
Period: Overall Study
Arm/Group | PD and F.A.D. Diagnostic Testing
Started | 62
Completed | 37
Not Completed | 25
Not completed — Lost to Follow-up | 10
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 6
Not completed — Unable to comply with study follow up | 2
Not completed — Investigator terminated participation | 1
Not completed — Insurance not covered | 2
Not completed — PD/FAD not done | 1

BASELINE CHARACTERISTICS:
Arm/Group | PD and F.A.D. Diagnostic Testing
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 61
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: Difference in Number of Magnetic Resonance Imaging (MRI)-Positive Discs Diagnosed Positive by Provocative Discography (PD) and Functional Anesthetic Discography (F.A.D.)
Description: For provocative discography (PD), a positive response at an individual disc requires all of the following findings: pain intensity (>=7/10 on 0-10 Numerical Rating Scale, NRS) as rated by subjects on injecting contrast into a disc; concordancy (pain reproduces typical back pain exactly). For Functional Anesthetic Discography (F.A.D.), a positive test at an individual disc level is defined as improvement in self-rated pain of >=2 Numerical Rating Scale (NRS) points AND >33% on 0-10 Numerical Rating Scale 10 minutes after injection of lidocaine.
Time Frame: Approximately 2 hours per subject
Population: Subjects which underwent Provocative Discography (PD) and Functional Anesthetic Discography (F.A.D.) consist of 1 population (N=50). Subjects which underwent either PD, F.A.D. or neither diagnostic test consist of a second population (all subjects enrolled, N=62). This is a diagnostic study. No imputation technique was used.
Measure: Number; unit: discs
Units Other Than Participants: discs
Arm/Group | PD and F.A.D. Diagnostic Testing
Number analyzed (Participants) | 50
Number analyzed (discs) | 66
discs
  PD - Negative and F.A.D. - Negative | 18
  PD - Negative and F.A.D. - Positive | 7
  PD - Positive and F.A.D. - Negative | 25
  PD - Positive and F.A.D. - Positive | 16
Statistical Analysis 1: Comparison: PD and F.A.D. Diagnostic Testing; Mcnemar test was used to test the difference between paired PD (provocative discography) and F.A.D. (Functional Anesthetic Discography) proportions; Test type: Superiority or Other; p = 0.002, McNemar; Exact test was used

ADVERSE EVENTS:
Arm/Group | PD and F.A.D. Diagnostic Testing
Serious Adverse Events (participants affected / at risk) | 1/62
Other Adverse Events (participants affected / at risk) | 10/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PD and F.A.D. Diagnostic Testing (N=62)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PD and F.A.D. Diagnostic Testing (N=62)
nausea (Gastrointestinal disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 2 (2)
back injury (Injury, poisoning and procedural complications) | 1 (1)
procedural pain (Injury, poisoning and procedural complications) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
monoparesis (Nervous system disorders) | 1 (1)
sciatica (Nervous system disorders) | 1 (1)
syncope vasovagal (Nervous system disorders) | 1 (1)
abnormal dreams (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
There were 12 subjects which did not undergo both PD (Provocative Discography) and F.A.D. (Functional Anesthetic Discography) and therefore could not be included in the primary endpoint analysis (analyzable population for primary endpoint = 50/62).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication, abstract, or presentation shall be submitted unless the multi-center report has been published. If report is not submitted within 24 months after completion, PI can present outcomes from their site. Proposed publications or presentations to be submitted to sponsor for review at least 60 days in advance. If proposed publication or presentation contains subject matter which is deemed to warrant intellectual property protection, sponsor may delay up to an additional 90 days.